CLINICAL TRIAL: NCT00409409
Title: A Randomised, Double-blind, Placebo-controlled, Multi-national, Multi-centre, Phase III Paediatric Study of the Efficacy and Safety of 300 IR Sublingual Immunotherapy (SLIT) Administered as Allergen-based Tablets Once Daily to Children Suffering From Grass Pollen Rhinoconjunctivitis
Brief Title: Efficacy and Safety of 300 IR Sublingual Immunotherapy (SLIT) Tablets in Children Suffering From Grass Pollen Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO52.06
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Allergy
Keywords: Sublingual immunotherapy; Grass pollen tablet; Allergic rhinoconjunctivitis
MeSH Terms: conditions — Hypersensitivity | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 300 IR (Experimental): 300 IR grass pollen allergen extract tablet
  Interventions: Drug: 300 IR grass pollen allergen extract tablet
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 300 IR grass pollen allergen extract tablet — One sublingual tablet daily during 4 months before pollen season and during pollen season
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR
Drug: Placebo tablet — One sublingual tablet daily during 4 months before pollen season and during pollen season
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
A phase III study to evaluate the efficacy and safety of SLIT for grass pollen allergens compared with placebo for reduction of symptoms and rescue medication usage in children.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 5 to 17 years.
* Written consent / assent.
* Grass pollen-related allergic rhinoconjunctivitis for at least the last two pollen seasons.
* Sensitised to grass pollen (positive SPT and grass pollen-specific IgE values of at least Class 2).
* Total symptom score on the Retrospective RTSS during the previous pollen season of greater than or equal to 12.

Exclusion Criteria:

* Patients who have received any desensitisation treatment for grass pollen.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2006-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Wahn, Professor, Principal Investigator — Charité - Campus Virchow Klinikum, Berlin, Germany
Locations (1):
- Charité - Campus Virchow Klinikum, Berlin, Germany

REFERENCES:
- [Result] Wahn U, Tabar A, Kuna P, Halken S, Montagut A, de Beaumont O, Le Gall M; SLIT Study Group. Efficacy and safety of 5-grass-pollen sublingual immunotherapy tablets in pediatric allergic rhinoconjunctivitis. J Allergy Clin Immunol. 2009 Jan;123(1):160-166.e3. doi: 10.1016/j.jaci.2008.10.009. Epub 2008 Nov 29. PMID 19046761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 16 DEC 2006, Last Patient Last Visit 12 SEP 2007
Period: Overall Study
Arm/Group | 300 IR | Placebo
Started | 139 | 139
Completed | 131 | 135
Not Completed | 8 | 4
Not completed — Adverse Event | 7 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Any other reason not above-mentioned | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all patients who received at least one dose of the investigational product and had a Retrospective Rhinoconjunctivitis Total Symptom Score (RRTSS) and at least one Rhinoconjunctivitis Total Symptom Score (RTSS) during the pollen period while on treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 IR | Placebo | Total
Number analyzed (Participants) | 131 | 135 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (3.34) | 11.2 (3.07) | 10.9 (3.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 95
  Male | 86 | 85 | 171

OUTCOME MEASURES:

1. Primary Outcome: Average Rhinoconjunctivitis Total Symptom Score (ARTSS)
Description: Average Rhinoconjunctivitis Total Symptom Score during the pollen period while participant on treatment.
  Participants assessed daily, during the pollen period, 6 rhinoconjunctivitis symptoms (sneezing, rhinorrhea, nasal pruritus, nasal congestion, ocular pruritus and watery eyes) each symptom is scored as follows: 0: no symptoms, 1: mild symptoms, 2: moderate symptoms, 3: severe symptoms. The sum of the 6 symptoms is the Rhinoconjunctivitis Total Symptom Score (RTSS) (range 0-18). The lower the score, the better the outcome.
Time Frame: Pollen period (average of 38.6 days)
Population: The Intent-to-treat (ITT) population included all patients who received at least one dose of the investigational product and had a Retrospective Rhinoconjunctivitis Total Symptom Score (RRTSS) and at least one Rhinoconjunctivitis Total Symptom Score (RTSS) in the pollen period while on treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale (range: 0 to 18)
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 131 | 135
Units on a scale (range: 0 to 18) | 3.25 (2.860) | 4.51 (2.931)
Statistical Analysis 1: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.0010, ANCOVA

ADVERSE EVENTS:
Time Frame: 4 months before the pollen period until the end of pollen period.
Description: Treatment-emergent Adverse Events (TEAEs) are defined as events that started on or after the first dose of the investigational product.
  Note: Serious Adverse Events and Other Adverse Events are described in Results Publication.
Arm/Group | 300 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 2/139 | 2/139
Other Adverse Events (participants affected / at risk) | 107/139 | 96/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=139) | Placebo (N=139)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
GASTRODUODENITIS (Gastrointestinal disorders) | 0 | 1
BURKITT'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=139) | Placebo (N=139)
COUGH (Respiratory, thoracic and mediastinal disorders) | 35 | 37
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 11 | 11
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 12 | 9
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 8 | 13
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 13 | 7
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 10
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 10 | 6
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 7 | 9
NASOPHARYNGITIS (Infections and infestations) | 19 | 18
PHARYNGITIS (Infections and infestations) | 6 | 16
TONSILLITIS (Infections and infestations) | 9 | 5
ORAL PRURITUS (Gastrointestinal disorders) | 46 | 6
OEDEMA MOUTH (Gastrointestinal disorders) | 18 | 0
HEADACHE (Nervous system disorders) | 11 | 24
EYE PRURITUS (Eye disorders) | 10 | 12
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 9
LIP SWELLING (Gastrointestinal disorders) | 7 | 1
CONJUNCTIVITIS (Eye disorders) | 4 | 7
LACRIMATION INCREASED (Eye disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No